CLINICAL TRIAL: NCT00644839
Title: A Phase 1, Open-Label, Fixed Sequence Study To Evaluate The Effect Of Multiple Dose Administration Of Omeprazole On The Single Dose Pharmacokinetics Of CP-945,598 In Healthy Overweight And Obese Subjects
Brief Title: Study Examing The Effect Of Omeprazole On Safety, Tolerability And How The Body Processes An Experimental Drug
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5351042
Record Dates: First submitted 2008-03-21; First posted 2008-03-27 (Estimated); Last update posted 2009-08-13 (Estimated); Status verified 2008-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CP-945,598 (Experimental)
  Interventions: Drug: CP-945,598

INTERVENTIONS:
Drug: CP-945,598 — Administration of CP-945,598 alone in period 1
Drug: CP-945,598 — Adminstration of CP-945,598 with omeprazole in period 2

SUMMARY:
Experiment in the test tube indicated that CP-945,598 becomes less soluble with increase of pH (less acidity). Changes in stomach acid levels may affect the solubility of CP-945,598, therefore, alters its availability in the blood. Omeprazole decreases acid levels in stomach. This study will compare the time course of drug concentrations in the body, safety, and tolerability of CP-945,598 given with and without omeprazole.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Body Mass Index (BMI) of 26.6 to 40.5 kg/m2.

Exclusion Criteria:

* Non-prescribed use of drugs or abuse of recreational drugs; recent treatment with experimental drugs or herbal experiments; EKG and blood pressure measurements falling outside of protocol-specified limits; history of regular alcohol or tobacco use exceeding protocol-specified limits; medically important health conditions; recent use of prescription or non-prescription medications.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2008-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Measurement of drug concentrations in serum from blood samples collected at 4 days before given omeprazole, and after second single dose of CP-945,598 on days 1-6, 8. | 1 day
Measurement of drug concentrations in serum from blood samples collected at various times after first single dose of CP-945,598 on days 1-6, 8, 15. | 1 day

SECONDARY OUTCOMES:
ECGs on the first and last day of the study | 2 days
Saftey laboratory tests (chemistry, hematology, urinalysis) on the first and last day of the study | 2 days
Vital signs (blood pressure, heart rate and respiratory rate) on the first and last day of the study | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Miami, Florida, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5351042&StudyName=Study%20Examing%20The%20Effect%20Of%20Omeprazole%20On%20Safety%2C%20Tolerability%20And%20How%20The%20Body%20Processes%20An%20Experimental%20Drug